CLINICAL TRIAL: NCT02499978
Title: Darunavir/Cobicistat and Dolutegravir to Maintain Virologic Suppression and Reduce NRTI-associated Toxicity (The 'deNUC' Study; TMC114HIV2030)
Brief Title: Darunavir/Cobicistat and Dolutegravir to Maintain Virologic Suppression and Reduce NRTI-associated Toxicity
Acronym: TMC114HIV2030
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry); University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Philip Grant, Assistant Professor of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: deNUC
Record Dates: First submitted 2015-07-14; First posted 2015-07-16 (Estimated); Last update posted 2021-07-09 (Actual); Status verified 2016-10

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — cobicistat mixture with darunavir; dolutegravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DRV/COBI, DTG Immediate switch (Experimental): DARUNAVIR/COBICISTAT (800mg/150MG), DOLUTEGRAVIR 50MG DAILY at randomization and follow through week 48.
  Interventions: Drug: Darunavir/Cobicistat; Drug: Dolutegravir
- DRV/COBI, DTG Delayed Switch (Active Comparator): DARUNAVIR/COBICISTAT (800MG150MG), DOLUTEGRAVIR 50MG DAILY at week 24 and follow through week 48.
  Interventions: Drug: Darunavir/Cobicistat; Drug: Dolutegravir

INTERVENTIONS:
Drug: Darunavir/Cobicistat — Fixed dose combination medication
  Other Names: Prezcobix, DRV/COBI
Drug: Dolutegravir — single tablet medication
  Other Names: Tivicay, DTG

SUMMARY:
This is a clinical research study to see if switching to Darunavir/Cobicistat ((PREZCOBIX™, DRV/COBI ) and Dolutegrivir (Tivicay®, DTG) in HIV-infected individuals with undetectable HIV viral load on nucleos(t)ide reverse transcriptase inhibitor (NRTI)-containing therapy will be effective in maintaining virologic suppression at 48 weeks of treatment.

DETAILED DESCRIPTION:
NRTIs have been a stalwart for treatment in both the pre- and post-ART eras. However, NRTIs have numerous toxicities partly due to the fact that they are analogs of naturally occurring nucleotides and interfere with the activity of numerous cellular functions. In highly treatment-experienced individuals with more than two active drugs in their salvage regimens, an NRTI-sparing regimen has been shown to be non-inferior to an NRTI-containing regimen [33]. However, studies with NRTI-sparing regimens not consisting of more than two active medications have generally been disappointing.

One limitation of earlier NRTI-sparing regimens has been a higher pill burden than more standard regimens. However, the approvals of DTG and the co-formulated DRV/COBI, both with well-established antiviral activities, may allow for a compact, effective, NRTI-sparing regimen. A switch to DTG/DRV/COBI in virologically suppressed HIV-infected individuals has the potential to avoid NRTI-associated toxicity while maintaining virologic suppression.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 infection, as documented by any licensed ELISA test kit and confirmed by Western blot at any time prior to study entry. A second antibody test by a method other than ELISA is acceptable as an alternative confirmatory test or a previous detectable HIV RNA level.

2 .Age ≥ 18 years

3. HIV-1 RNA <50 copies/mL while on a stable antiretroviral regimen for at least 6 months prior to study entry excluding blips (i.e., a single measurement <200 copies/mL preceded and followed by measurements <50 copies/mL)

4. At screening, patient on a stable antiretroviral regimen containing at least one NRTI and a PI, NNRTI, or INSTI

5. No changes in antiretroviral regimen in the six months prior to screening (except for a switch to a coformulated tablet from the component tablets)

6. A desire to switch off current antiretroviral therapy due to: a) Renal dysfunction (microalbuminuria/proteinuria or CrCl<70 mL/min/1.73 m2) on tenofovir disoproxil fumarate (TDF) of tenofovir al; b) Osteopenia or osteoporosis on a TDF-containing regimen (i.e., lowest T-score ≥1.0 standard deviation below the young adult mean measured by dual-energy x-ray absorptiometry); c) Peripheral neuropathy or lipoatrophy at least partially attributable to ongoing NRTI use; d) Intermediate or high Framingham risk (i.e., ≥10% 10-year risk) on an abacavir-containing regimen; e) Patient preference.

7. Laboratory values within six months of screening visit

* Hemoglobin ≥8.0 g/dL
* Platelet count ≥40,000/mm3
* AST, ALT, and alkaline phosphatase ≤5 × ULN
* Total bilirubin ≤2.5 x ULN (except for those on atazanavir-containing regimens)
* Calculated creatinine clearance (CrCl) ≥45 mL/min as estimated by the Cockcroft-Gault equation:

For men, (140 - age in years) x (body weight in kg) ÷ (serum creatinine in mg/dL x 72) = CrCl (mL/min)*

*For women, multiply the result by 0.85 = CrCl (mL/min)

8. For women of reproductive potential, negative serum or urine pregnancy test at screening and a negative urine pregnancy test at the entry visit prior to randomization and also agreeable to using a contraceptive of choice during the study period.

"Women of reproductive potential" are defined as women who have not been post-menopausal for at least 24 consecutive months (i.e., who have had menses within the preceding 24 months) and have not undergone surgical sterilization (i.e., hysterectomy, bilateral oophorectomy, or tubal ligation)

Exclusion Criteria:

1. Current CD4+ T-cell count <200 cells/µL
2. Current antiretroviral regimen consisting of three of more antiretroviral classes
3. History of genotypic resistance, phenotypic resistance or intolerance to either DRV or DTG.

   Prohibited protease mutations: V11I, V32I, L33F, I47V/A/L, I50V, I54T/S/L/M, T74P, L76V, V82F, I84V, or L89V

   Prohibited INSTI mutations: E92Q, E92K/A, G140S/A/C, Q148H/R/K or Q148 substitution plus any of the following: L74I/M, E138A/D/K/T, G140A/S, Y143H/R, E157Q, G163E/K/Q/R/S, or G193E/R.
4. History of virologic failure while on an INSTI prior to study enrollment
5. Severe hepatic impairment (Child Pugh Class C)
6. Hepatitis B Surface Antigen Positive
7. Breastfeeding, pregnancy, or plans to become pregnant during the study
8. Known allergy/sensitivity to any study drug or their formulations.
9. Receipt or planned receipt of prohibited concomitant medications (See section 5.2.1)
10. Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study procedures and treatment.
11. Serious medical illness that, in the opinion of the site investigator, precludes safe participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-05; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Virologic suppression (24 weeks) | 24 weeks
  Compare between arms the proportion of patients maintaining virologic suppression (i.e., no confirmed HIV RNA levels ≥200 copies/mL) at Week 24

SECONDARY OUTCOMES:
Virologic Suppression (48 weeks) | 48 weeks
  Evaluate the proportion of participants who maintain virologic suppression 24 weeks post-switch (i.e. at 24 weeks in the immediate switch arm and at 48 weeks in the delayed switch arm)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Grant, MD, Study Director — Stanford University; Sean Collins, MD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Stanford Univerity, Stanford, California
  - University of Colorado, Aurora, Colorado